CLINICAL TRIAL: NCT04637737
Title: Effect of Anterioposterior Weight Shifting Training With Visual Biofeedback in Subacute Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0383
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental)
  Interventions: Device: anterioposterior Weight Shifting Training with Visual Biofeedback
- Control group (Other)
  Interventions: Behavioral: Conventional therapy

INTERVENTIONS:
Device: anterioposterior Weight Shifting Training with Visual Biofeedback — The training group received an additional anterioposterior weight shifting training with visual Biofeedback 5 times per week for 4weeks. AP training is made to instantly know your training status during training by measuring and processing the foot pressure in real time using the F-Scan (Tekscan) hardware system and Software Development Kit (SDK).
  Before training, all patients are instructed to place both feet at shoulder width, place the inverted foot approximately 30 cm in front of the unaffected side foot, move the body forward with the chest straight in an upright position, and be instructed to put the weight on the affected side.
  On the screen shown, measure the maximum weight distribution during the first 10 times and set the value added by 5% as the target value.
  It is designed to induce the maximum weight shift through the archery game.
  Arms: Training group
Behavioral: Conventional therapy — The control group received the usual gait training.
  Arms: Control group

SUMMARY:
Asymmetric gait patterns of stroke is one of the most important functional activities to enable community participation, it is major goal for stroke patients. Reported that the stroke patients had asymmetry at stance time, single stance, double support time, and swing time compared to normal people, and claimed that the most important factor was step length. According to Albert et al., patients with an asymmetric gait pattern have a long double support phase and a healthy side single support phase, and less weight shift to the affected side. Recent studies have shown that visual feedback for weight shift may be helpful to obtain a symmetrical posture after stroke. However, no study has been conducted on the therapeutic effect on gait asymmetry and patterns. We aimed to investigate the effect of Anterioposterior Weight Shifting Training with Visual Biofeedback in subacute post-stroke patients on gait asymmetry and pattern.

40 subacute post-stroke patients with Step Length Asymmetry were enrolled in this study. The subjects were randomly assigned into two groups. The training group received an additional anterioposterior weight shifting training with visual Biofeedback 5 times per week for 4weeks. The control group received the usual gait training. The spatiotemporal and kinematic data were obtained during walking through 3D motion analysis. Functional Ambulation Category, Self-selected walking speed, Maximum safe walking speed, Berg balance Test (BBT), Fugl-Meyer Assessment (FMA), Medical Research Council Score (MRC), Functional Independent Measure-mobility, Timed Up and Go test (TUG) were assessed at pre, during, post- training, and 4week follow-up. Those were compared between two groups by repeated measures ANOVA.

ELIGIBILITY:
Inclusion Criteria:

1. less than 6 months after onset of the stroke
2. can stand and walk independently 10m
3. K-MMSE score of at least 15
4. have asymmetrical gait pattern with Step length asymmetric ratio greater than 1.1
5. over 20 years of age.

Exclusion Criteria:

1. quadriplegia
2. past history of stroke
3. past history of Musculoskeletal disease or history of Neurological diseases

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-10-01; Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Step Length Asymmetric Ratio | before training(0week)
  Step Length Asymmetric Ratio = paretic step length/non paretic step length
Step Length Asymmetric Ratio | during training(2week)
  Step Length Asymmetric Ratio = paretic step length/non paretic step length
Step Length Asymmetric Ratio | after training(4week)
  Step Length Asymmetric Ratio = paretic step length/non paretic step length
Step Length Asymmetric Ratio | Follow up(8week)
  Step Length Asymmetric Ratio = paretic step length/non paretic step length
Step Length Asymmetric Index | before training(0week)
  Step Length Asymmetric Index = paretic step length-non paretic step length/0.5[paretic step length +non paretic step length]
Step Length Asymmetric Index | during training(2week)
  Step Length Asymmetric Index = paretic step length-non paretic step length/0.5[paretic step length +non paretic step length]
Step Length Asymmetric Index | after training(4week)
  Step Length Asymmetric Index = paretic step length-non paretic step length/0.5[paretic step length +non paretic step length]
Step Length Asymmetric Index | Follow up(8week)
  Step Length Asymmetric Index = paretic step length-non paretic step length/0.5[paretic step length +non paretic step length]

CONTACTS AND LOCATIONS:
Overall Officials: Deog Young Kim, Principal Investigator — Severance Hospital
Locations (1):
- Department and Research Institute of Rehabilitation Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No